CLINICAL TRIAL: NCT00261768
Title: Efficacy of Digital Noise Reduction Strategies: A Hearing Aid Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Wilson, Richard - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3011R
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Sensorineural Hearing Loss
Keywords: Aging; hearing aids; hearing loss, sensorineural; speech recognition
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Noise reduction on
  Interventions: Behavioral: Digital noise reduction

INTERVENTIONS:
Behavioral: Digital noise reduction

SUMMARY:
The purpose of this study is to see if noise reduction programs in digital hearing aids help patients hear better than hearing aids without these programs. We also want to know if we can predict how successful patients will be with hearing aids.

DETAILED DESCRIPTION:
The first goal of this project is to examine the efficacy of digital hearing aids incorporating three noise reduction strategies (i.e., directional microphones alone vs. directional microphones with DSP noise reduction algorithm 1 vs. directional microphones with DSP noise reduction algorithm 2) in terms of both speech understanding outcomes and functional outcomes. The second goal is to identify individual characteristics that are predictive of successful functional outcomes with hearing aids.

This study employs a multi-site, randomized, blinded, 2x2 factorial parallel group design. Three hundred subjects will be studied at three VA Medical Centers (Mountain Home, TN; Bay Pines, FL; and Los Angeles, CA) over a period of three years.

Objective (word recognition ability and performance with degraded speech stimuli) subjective (self-assessment questionnaires, personality and depression assessments) and cost-effectiveness assessments will be measured for 4 randomized treatment groups receiving different digital hearing aid technology. Subjects will be randomly assigned to wear hearing aids with directional microphones alone or directional microphones with noise reduction algorithm 1 or directional microphones with noise reduction algorithm 2 for a period of 8 weeks. Subjects will complete post-testing after 8 weeks of hearing aid use.

ELIGIBILITY:
Inclusion Criteria:

1. adult onset sensorineural hearing loss
2. English as the first language
3. bilateral symmetrical sensorineural hearing loss
4. Patient is a candidate for directional microphone technology.
5. average audiometric thresholds for 500, 1000, 2000, 3000, and 4000 Hz no better than 25-dB HL in either ear.
6. no history of hearing aid use in the past 10 years
7. appropriate cognitive skills to participate in the study as determined by a passing score on the Mini Mental Scale.
8. Patient has a local telephone and address.

Exclusion Criteria:

1. evidence of outer ear, middle ear, or retrocochlear pathology
2. any threshold from 500 to 2000 Hz exceeds 70-dB HL
3. known neurological or psychiatric disorders as determined by chart review
4. known comorbid diseases that would prevent completion of the study as determined by chart review
5. visual impairment that would interfere with reading the questionnaires

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Words in Noise Test | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wilson, PhD, Principal Investigator — James H. Quillen VA Medical Center
Locations (2):
- United States (2):
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - James H. Quillen VA Medical Center, Mountain Home, Tennessee